CLINICAL TRIAL: NCT00424307
Title: Development of Auditory Skills in Young Deaf Children With Bilateral Cochlear Implants
Brief Title: Bilateral Cochlear Implant Benefit in Young Children
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Advanced Bionics (Industry)
Responsible Party: Kenneth Ripley, Advanced Bionics, LLC
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ACR0906
Record Dates: First submitted 2007-01-17; First posted 2007-01-19 (Estimated); Last update posted 2011-06-27 (Estimated); Status verified 2011-06

CONDITIONS: Hearing Loss
MeSH Terms: conditions — Hearing Loss

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Device: HiResolution Bionic Ear System

SUMMARY:
The primary purpose of this study is to track patient outcomes for bilateral cochlear implant recipients in a cohort of 60 children, ages 12 to 36 months at time of surgery, who receive two implants in the same operation or in two different surgeries with the initial fitting of the devices separated by no more than six months.

ELIGIBILITY:
Inclusion Criteria:

* Profound bilateral hearing loss
* Have independently elected to undergo bilateral implantation of Advanced Bionics HiResolution Bionic Ear System
* Age at implant: 12-36 months
* No previous cochlear implant use
* English as the primary language spoken in the home
* Parental willingness to follow study protocol

Exclusion Criteria:

* Deafness secondary to meningitis
* Presence of other conditions that could affect study participation

Ages: 12 Months to 36 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 60 (Estimated)
Dates: Start 2007-01; Primary Completion 2012-04 (Estimated); Study Completion 2012-04 (Estimated)

PRIMARY OUTCOMES:
Assessment of Speech Perception Skills | Various time points

SECONDARY OUTCOMES:
Health-Related Quality of Life and Assessment of Communicative Performance | Various time points

CONTACTS AND LOCATIONS:
Overall Officials: Mary Joe Osberger, Ph.D., Study Chair — Advanced Bionics
Locations (14):
- United States (13):
  - Children's HEAR Center, Birmingham, Alabama
  - House Ear Institute, Los Angeles, California
  - University of California, San Francisco, San Francisco, California
  - Tampa Bay Hearing and Balance Center, Tampa, Florida
  - The Children's Memorial Hospital, Chicago, Illinois
  - Carle Foundation Hospital, Urbana, Illinois
  - Massachusetts Eye and Ear Infirmary, Boston, Massachusetts
  - Spectrum Health Hospital, Grand Rapids, Michigan
  - Midwest Ear Institute, Kansas City, Missouri
  - Washington University of St. Louis, St Louis, Missouri
  - Boys Town National Research Hospital, Omaha, Nebraska
  - New York University, New York, New York
  - Dallas Otolaryngology Associates, Dallas, Texas
- Glenrose Rehab Hospital, Edmonton, Alberta, Canada